CLINICAL TRIAL: NCT03856931
Title: Behaviours and Emotions in Preschoolers - Detecting Mental Health Problems in Preschool Children in a Primary Care Population
Brief Title: Behaviours and Emotions in Preschoolers
Acronym: BeEPS
Status: Completed | Type: Observational
Sponsor: TARGetKids! (Other)
Collaborators: The Hospital for Sick Children (Other); Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Alice Charach, Staff Psychiatrist, The Hospital for Sick Children
Other Study IDs: 1000056960
Record Dates: First submitted 2019-02-26; First posted 2019-02-27 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Mental Health Wellness; Emotional Problem; Behavioural Problem; Post Partum Depression
Keywords: mental health; preschool; SDQ; parental depression
MeSH Terms: conditions — Mental Disorders; Depression, Postpartum; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this TARGet Kids! Study, we want to find out whether a short questionnaire can be used to help find out about mental health problems in preschool age children.

DETAILED DESCRIPTION:
Research indicates that more than 1 in 10 preschoolers have significant social, emotional and behavioural problems also known as mental health problems. Unfortunately, parents and doctors rarely identify mental health problems in young children in order to begin treatment. We are testing a short five-minute questionnaire completed by parents to see if this may help a doctor notice if a child has social, emotional and behavioural problems.

In addition, we also hope to find out if the presence of feelings of stress and depression in on or both parents may be associated with mental health problems in their preschool child.

This study is being conducted by researchers at SickKids and St. Michael's Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Child is between age 2 to 4 years.
2. Parent is the primary caretaker for the child and is able to speak, read and understand English well enough to complete the forms and the PAPA interview.
3. Either one or both parents (primary caretakers) are available to participate in the study.

Exclusion Criteria:

1. Children with associated health conditions affecting growth (e.g. failure to thrive, cystic fibrosis);
2. Children with any acute or chronic conditions except for asthma and high functioning autism;
3. Children with severe developmental delay;
4. Children with a gestational age of less than 32 weeks;
5. Families who are not fluent in English.

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: TARGet Kids! (The Applied Research Group for Kids) is a research project enrolling healthy children aged 0-5 years during their primary-care health supervision visits with their primary care physician who is a Community Physician Collaborator with the TARGetKids! primary-care practice-based research network. The BeEPS study will recruit participants from within the TARGet Kids! cohort.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Total difficulties score | 3 months
  As measured by the preschool strengths and difficulties questionnaire (P-SDQ)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Charach, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided